CLINICAL TRIAL: NCT01309256
Title: Multi-institutional Study on the Assessment of Robotic Surgery for Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2010-0659
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Gastric Cancer
Keywords: distal gastrectomy; Robotic gastrectomy; registry; learning curve; cost-effectiveness; quality of life; acute inflammatory reaction; Robotic and laparoscopic surgery
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- R-robot group: retrospective robot group
- P-robot group: prospective robot group
- P-laparoscopic group: prospective laparoscopic group

SUMMARY:
Minimally invasive surgery revolutionized the field of gastric cancer surgery. The surgical robot was introduced to alleviate the difficulty of laparoscopic surgery. Although many studies have reported successful outcomes for robotic surgery, there is no multicenter prospective analysis regarding the advantage of the robotic gastrectomy. The aim of this study is to analyze the surgical outcomes of the robotic gastrectomy focusing on the learning curve, cost-effectiveness, quality of life, and acute-inflammatory reaction in comparison with laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria for prospective study participants

* Patients must have documented diagnosis of gastric cancer
* Patients receiving laparoscopic gastric cancer surgery without preoperative evidence of serosal invasion and distant lymph node metastasis as determined by preoperative CT-scan, upper endoscopy, and endoscopic ultrasound.
* Patients who have received comprehensive explanation about the planned study, understand and accept all the terms of the study and willingly give consent to participate in all the required elements of the study

Inclusion Criteria for retrospective study participants

- Any patients who underwent robotic gastrectomy in Korea

Exclusion Criteria for prospective study participants

* Patients without mental competence
* Patients who are illiterate
* Patients who are pregnant
* Patients < 20 years old

Exclusion Criteria for retrospective study participants

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Registration of all robotic gastrectomies performed in South Korea | at the end of the study
Learning curve (operation time and surgical outcome) of robotic gastrectomy | from the start of the operation to discharge of the patient (usually two weeks after the operation)
Cost-effectiveness comparison between robotic and laparoscopic gastrectomy | from admission to discharge of the patient (usually from two days before the operation until two weeks after the operation)
Quality of life after robotic and laparoscopic gastrectomy | One day before operation, first OPD visit after the operation (two weeks after the operation), 3M, 12M, 36M, and 60M after the operation
Acute-inflammatory response after undergoing robotic and laparoscopic gastrectomy | preop, 2hr, 24hr, 4days and 30 days after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Song J, Oh SJ, Kang WH, Hyung WJ, Choi SH, Noh SH. Robot-assisted gastrectomy with lymph node dissection for gastric cancer: lessons learned from an initial 100 consecutive procedures. Ann Surg. 2009 Jun;249(6):927-32. doi: 10.1097/01.sla.0000351688.64999.73. PMID 19474671
- [Background] Song J, Kang WH, Oh SJ, Hyung WJ, Choi SH, Noh SH. Role of robotic gastrectomy using da Vinci system compared with laparoscopic gastrectomy: initial experience of 20 consecutive cases. Surg Endosc. 2009 Jun;23(6):1204-11. doi: 10.1007/s00464-009-0351-4. Epub 2009 Mar 5. PMID 19263147
- [Background] Kim MC, Heo GU, Jung GJ. Robotic gastrectomy for gastric cancer: surgical techniques and clinical merits. Surg Endosc. 2010 Mar;24(3):610-5. doi: 10.1007/s00464-009-0618-9. Epub 2009 Aug 18. PMID 19688399
- [Background] Song J, Lee HJ, Cho GS, Han SU, Kim MC, Ryu SW, Kim W, Song KY, Kim HH, Hyung WJ; Korean Laparoscopic Gastrointestinal Surgery Study (KLASS) Group. Recurrence following laparoscopy-assisted gastrectomy for gastric cancer: a multicenter retrospective analysis of 1,417 patients. Ann Surg Oncol. 2010 Jul;17(7):1777-86. doi: 10.1245/s10434-010-0932-4. Epub 2010 Feb 12. PMID 20151217
- [Background] Lee HJ, Kim HH, Kim MC, Ryu SY, Kim W, Song KY, Cho GS, Han SU, Hyung WJ, Ryu SW; Korean Laparoscopic Gastrointestinal Surgery Study Group. The impact of a high body mass index on laparoscopy assisted gastrectomy for gastric cancer. Surg Endosc. 2009 Nov;23(11):2473-9. doi: 10.1007/s00464-009-0419-1. Epub 2009 Apr 3. PMID 19343439
- [Background] Kim MC, Kim W, Kim HH, Ryu SW, Ryu SY, Song KY, Lee HJ, Cho GS, Han SU, Hyung WJ; Korean Laparoscopic Gastrointestinal Surgery Study (KLASS) Group. Risk factors associated with complication following laparoscopy-assisted gastrectomy for gastric cancer: a large-scale korean multicenter study. Ann Surg Oncol. 2008 Oct;15(10):2692-700. doi: 10.1245/s10434-008-0075-z. Epub 2008 Jul 29. PMID 18663532
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Derived] Kim MS, Kim WJ, Hyung WJ, Kim HI, Han SU, Kim YW, Ryu KW, Park S. Comprehensive Learning Curve of Robotic Surgery: Discovery From a Multicenter Prospective Trial of Robotic Gastrectomy. Ann Surg. 2021 May 1;273(5):949-956. doi: 10.1097/SLA.0000000000003583. PMID 31503017
- [Derived] Kim HI, Han SU, Yang HK, Kim YW, Lee HJ, Ryu KW, Park JM, An JY, Kim MC, Park S, Song KY, Oh SJ, Kong SH, Suh BJ, Yang DH, Ha TK, Kim YN, Hyung WJ. Multicenter Prospective Comparative Study of Robotic Versus Laparoscopic Gastrectomy for Gastric Adenocarcinoma. Ann Surg. 2016 Jan;263(1):103-9. doi: 10.1097/SLA.0000000000001249. PMID 26020107